CLINICAL TRIAL: NCT00801398
Title: An Open-Label, Ascending, Two-Part, Single- and Multiple-Dose Evaluation of the Safety, Pharmacokinetics, and Effectiveness of Oxymorphone for Acute Postoperatiave Pain in Pediatric Subjects
Brief Title: Open-Label Safety and Tolerability Study of Oxymorphone for Acute Postoperative Pain in Pediatric Subjects.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EN3203-010
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2018-12

CONDITIONS: Postoperative Pain
Keywords: Opioid tolerant; Pediatric; Pain; Non malignant; Malignant
MeSH Terms: conditions — Pain, Postoperative; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Oxymorphone IR (Experimental): Open-Label, 2 part ascending-dose multicenter study
  Interventions: Drug: Oxymorphone IR

INTERVENTIONS:
Drug: Oxymorphone IR — Open-label, 2 part, ascending dose, single and multiple dose q4-6 hrs up to 48 hrs
  Other Names: Opana IR

SUMMARY:
When post-operative parenteral analgesia is discontinued, oral dosing with study medication may begin once the subject has developed a moderate level of pain as defined by a 100 mm VAS (pain intensity score greater than or equal to 40).

This post marketing study was required by the FDA. Endo Pharmaceuticals Inc. no longer promotes opioids and no longer markets Opana® ER.

ELIGIBILITY:
Inclusion Criteria:

* Male or female > 12 to 17 years of age, inclusive
* Weigh at least 50 kg
* Postoperative oral opioid analgesia required for at least 24 hours or 48 hours following postoperataive parenteral analgesia
* Are expected to be hospitalized for the duration of the study

Exclusion Criteria:

* Known allergy to, or a significant reaction to, oxymorphone or another opioid
* Life expectancy of < 4 weeks
* Positive pregnancy test at screening

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 58 (Actual)
Dates: Start 2009-02-17 (Actual); Primary Completion 2011-04-18 (Actual); Study Completion 2011-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Endo Pharmaceuticals
Locations (11):
- United States (11):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Stanford University School of Medicine, Stanford, California
  - The Children's Hospital, Aurora, Colorado
  - Children's Research Institute, Washington D.C., District of Columbia
  - St. Joseph's Children's Hospital of Tampa, Tampa, Florida
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Monroe Carell Jr. Children's Hospital at Vanderbilt, Nashville, Tennessee
  - University of Texas Southwestern Medical Center at Dallas, Dallas, Texas
  - University of Washington, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Multiple Dose of Oxymorphone: 5mg Tablet | Multiple Dose of Oxymorphone IR: 10mg Tablet | Multiple Dose of Oxymorphone IR: 15mg Tablet
Started | 13 | 9 | 11 | 9 | 8 | 8
Completed | 7 | 0 | 4 | 3 | 1 | 5
Not Completed | 6 | 9 | 7 | 6 | 7 | 3

BASELINE CHARACTERISTICS:
Population: ITT Population; Single Dose Total = 33; Multiple Dose Total = 25;
Groups:
- Total: Total of all reporting groups
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Multiple Dose of Oxymorphone IR: 5mg Tablet | Multiple Dose of Oxymorphone IR: 10mg Tablet | Multiple Dose of Oxymorphone IR: 15mg Tablet | Total
Number analyzed (Participants) | 13 | 9 | 11 | 9 | 8 | 8 | 58
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Single Dose of Oxymorphone IR Overall (N=33): Mean 14.9 SD (1.64) Multiple Dose of Oxymorphone IR Overall (N=25): Mean 15.2 SD (1.13)
  years | 14.9 (1.71) | 15.3 (1.66) | 14.6 (1.63) | 15.0 (0.71) | 15.3 (1.58) | 15.5 (1.07) | 15.07 (1.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 8 | 4 | 6 | 4 | 38
  Male | 4 | 2 | 3 | 5 | 2 | 4 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 2 | 0 | 1 | 3
  Not Hispanic or Latino | 13 | 9 | 11 | 7 | 8 | 7 | 55
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 1 | 0 | 1 | 0 | 6
  White | 11 | 7 | 10 | 9 | 7 | 6 | 50
  More than one race | 0 | 0 | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13 | 9 | 11 | 9 | 8 | 8 | 58

OUTCOME MEASURES:

1. Primary Outcome: Summary of Visual Analog Scales (VAS) of Pain Intensity Change From Baseline by Treatment Group With Single Dose of Oxymorphone IR Tablet and Multiple Dose of Oxymorphone IR Tablet
Description: Change from Baseline in 100-mm Visual Analog Scales (VAS) in Multiple Dose of Oxymorphone IR Tablet
Time Frame: Single Dose Timeframe: 15min, 30min, 1h, 2h, 3h, 4h, 6h or Rescue; Multiple Dose Timeframe: 15min, 30min, 1h, 2h, 3h, 4h, 6h, subsequent doses every 4-6 hours (Multiple Dose #1-11), and Early Termination
Population: ITT Population
Measure: Mean (Standard Deviation); unit: mm
Groups:
- Change From Baseline Single Dose of Oxymorphone IR: 5mg Tablet; Change From Baseline Single Dose Oxymorphone IR: 10mg Tablet; Change From Baseline Single Dose Oxymorphone IR: 15mg Tablet; Change From Baseline Multiple Dose Oxymorphone IR: 5mg Tablet; Change From Baseline Multiple Dose Oxymorphone IR: 10mg Tablet; Change From Baseline Multiple Dose Oxymorphone IR: 15mg Tablet: Change from Baseline
Arm/Group | Change From Baseline Single Dose of Oxymorphone IR: 5mg Tablet | Change From Baseline Single Dose Oxymorphone IR: 10mg Tablet | Change From Baseline Single Dose Oxymorphone IR: 15mg Tablet | Change From Baseline Multiple Dose Oxymorphone IR: 5mg Tablet | Change From Baseline Multiple Dose Oxymorphone IR: 10mg Tablet | Change From Baseline Multiple Dose Oxymorphone IR: 15mg Tablet
Number analyzed (Participants) | 13 | 9 | 11 | 9 | 8 | 8
mm
  15 Minutes Post Dose/ 15 Minutes Post First Dose: number analyzed (Participants) | 13 | 9 | 10 | 9 | 8 | 7
  15 Minutes Post Dose/ 15 Minutes Post First Dose | -13.4 (22.86) | -22.2 (17.79) | -21.6 (13.59) | -16.7 (23.31) | 0.5 (9.56) | -17.4 (13.46)
  30 Minutes Post Dose/30 Minutes Post First Dose: number analyzed (Participants) | 13 | 9 | 10 | 9 | 8 | 8
  30 Minutes Post Dose/30 Minutes Post First Dose | -12.8 (36.90) | -13.7 (28.32) | -22.9 (19.87) | -18.3 (25.84) | 3.1 (22.33) | -23.0 (15.94)
  1 Hour Post Dose/1 Hour Post First Dose: number analyzed (Participants) | 13 | 8 | 10 | 8 | 6 | 8
  1 Hour Post Dose/1 Hour Post First Dose | -24.70 (36.74) | -17.4 (28.64) | -29.8 (20.02) | -22.0 (25.13) | -7.8 (18.90) | -28.3 (15.00)
  2 Hours Post Dose/2 Hours Post First Dose: number analyzed (Participants) | 12 | 4 | 9 | 8 | 4 | 8
  2 Hours Post Dose/2 Hours Post First Dose | -19.3 (29.07) | -29.0 (25.55) | -33.8 (20.10) | -14.4 (36.56) | -6.3 (22.04) | -12.9 (34.37)
  3 Hours Post Dose/3 Hours Post First Dose: number analyzed (Participants) | 10 | 3 | 8 | 4 | 4 | 6
  3 Hours Post Dose/3 Hours Post First Dose | -35.4 (26.97) | -29.3 (20.21) | -28.6 (16.75) | -25.8 (40.17) | -15.5 (19.67) | -24.7 (20.70)
  4 Hours Post Dose/4 Hours Post First Dose: number analyzed (Participants) | 9 | 2 | 4 | 5 | 4 | 6
  4 Hours Post Dose/4 Hours Post First Dose | -36.2 (25.03) | -19.5 (45.96) | -31.5 (14.20) | -34.8 (31.65) | -7.5 (29.33) | -10.8 (20.64)
  6 Hrs Post Dose or Rescue/6 Hours Post First Dose: number analyzed (Participants) | 7 | 5 | 6 | 1 | 3 | 3
  6 Hrs Post Dose or Rescue/6 Hours Post First Dose | -34.4 (25.32) | -3.0 (21.85) | -18.2 (18.73) | -41.0 (NA) — SD cannot be derived based on one subject data point | -6.0 (20.22) | -38.3 (9.45)
  Multiple Dose #1: number analyzed (Participants) | 0 | 0 | 0 | 3 | 4 | 5
  Multiple Dose #1 |  |  |  | -28.0 (14.11) | -15.0 (17.72) | -25.2 (11.65)
  Multiple Dose #2: number analyzed (Participants) | 0 | 0 | 0 | 2 | 4 | 5
  Multiple Dose #2 |  |  |  | -33.5 (10.61) | 0.8 (7.04) | -17.6 (20.70)
  Multiple Dose #3: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5
  Multiple Dose #3 |  |  |  | -33.5 (10.61) | 4.0 (18.38) | -26.4 (12.38)
  Multiple Dose #4: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5
  Multiple Dose #4 |  |  |  | -33.0 (11.31) | 18.5 (13.44) | -25.4 (4.04)
  Multiple Dose #5: number analyzed (Participants) | 0 | 0 | 0 | 2 | 2 | 5
  Multiple Dose #5 |  |  |  | -38.0 (4.24) | -19.0 (41.01) | -21.6 (19.03)
  Multiple Dose #6: number analyzed (Participants) | 0 | 0 | 0 | 2 | 1 | 5
  Multiple Dose #6 |  |  |  | -38.0 (4.24) | -1.0 (NA) — SD cannot be derived based on one subject data point | -32.8 (15.32)
  Multiple Dose #7: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 5
  Multiple Dose #7 |  |  |  | -33.0 (NA) — SD cannot be derived based on one subject data point | -36.0 (NA) — SD cannot be derived based on one subject data point | -26.6 (21.80)
  Multiple Dose #8: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 3
  Multiple Dose #8 |  |  |  | -35.0 (NA) — SD cannot be derived based on one subject data point | -8.0 (NA) — SD cannot be derived based on one subject data point | -32.7 (13.65)
  Multiple Dose #9: number analyzed (Participants) | 0 | 0 | 0 | 1 | 1 | 3
  Multiple Dose #9 |  |  |  | -34.0 (NA) — SD cannot be derived based on one subject data point | -6.0 (NA) — SD cannot be derived based on one subject data point | -22.7 (15.50)
  Multiple Dose #10: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 3
  Multiple Dose #10 |  |  |  |  | -6.0 | -29.0 (17.06)
  Multiple Dose #11: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 1
  Multiple Dose #11 |  |  |  |  | -29.0 (NA) — SD cannot be derived based on one subject data point | -17.0 (NA) — SD cannot be derived based on one subject data point
  Early Termination: number analyzed (Participants) | 0 | 0 | 0 | 4 | 5 | 0
  Early Termination |  |  |  | 1.8 (50.74) | 7.4 (42.29) |

2. Primary Outcome: Subjects Taking Rescue Medication
Description: Percentages are based on the number of subjects in each treatment group.
Time Frame: first dose through 48 hours after first dose
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Single Dose of Oxymorphone IR: 5mg Tablet; Single Dose of Oxymorphone IR: 10mg Tablet; Single Dose of Oxymorphone IR: 15mg Tablet; Multiple Dose of Oxymorphone: 5mg Tablet; Multiple Dose of Oxymorphone IR: 10mg Tablet; Multiple Dose of Oxymorphone IR: 15mg Tablet: Subjects With at Least One Rescue Medication
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Multiple Dose of Oxymorphone: 5mg Tablet | Multiple Dose of Oxymorphone IR: 10mg Tablet | Multiple Dose of Oxymorphone IR: 15mg Tablet
Number analyzed (Participants) | 13 | 9 | 11 | 9 | 8 | 8
Participants | 9 | 9 | 7 | 5 | 6 | 4

3. Secondary Outcome: AUC(0-t) of Single Dose of Oxymorphone by Treatment Group
Description: AUC0-t: Area under the concentration versus time curve from time 0 to the last measured concentration (Ct), calculated by linear trapezoidal rule
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | 6-OH-Oxymorphone (ng/mL): 10mg | 6-OH-Oxymorphone (ng/mL): 15mg
Number analyzed (Participants) | 9 | 6 | 9 | 8 | 6 | 9
ng*hr/mL | 6.395 (6.0752) | 3.766 (2.2587) | 67.040 (150.7979) | 1.544 (1.8794) | 3.040 (1.1625) | 7.354 (3.3255)

4. Secondary Outcome: AUC(0-inf) of Single Dose of Oxymorphone by Treatment Group
Description: AUC0-inf: Area under the concentration versus time curve from time 0 to infinity, calculated as AUC0-t + Ct/terminal rate constant (single-dose period only), where Ct is the concentration at the time of the last quantifiable concentration
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | Single Dose of 6-OH-Oxymorphone: 10mg Tablet | Single Dose 6-OH-Oxymorphone: 15mg Tablet
Number analyzed (Participants) | 9 | 3 | 8 | 5 | 5 | 9
ng*hr/mL | 7.632 (6.6828) | 10.223 (6.5195) | 109.294 (257.5421) | 4.987 (7.5732) | 8.692 (10.2430) | 12.795 (8.8385)

5. Secondary Outcome: Cmax of Single Dose of Oxymorphone by Treatment Group
Description: Cmax: Maximum plasma concentration; the highest concentration observed during a dosage interval
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | Single Dose of 6-OH-Oxymorphone: 10mg Tablet | Single Dose 6-OH-Oxymorphone: 15mg Tablet
Number analyzed (Participants) | 9 | 6 | 9 | 8 | 6 | 9
ng/mL | 1.243 (1.2192) | 0.828 (0.6892) | 5.295 (10.6386) | 0.314 (0.3276) | 0.487 (0.2853) | 0.940 (0.5212)

6. Secondary Outcome: Tmax of Single Dose of Oxymorphone by Treatment Group
Description: Tmax: The time at which Cmax was observed
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | Single Dose of 6-OH-Oxymorphone: 10mg Tablet | Single Dose 6-OH-Oxymorphone: 15mg Tablet
Number analyzed (Participants) | 9 | 6 | 9 | 8 | 6 | 9
hour | 4.898 (3.9645) | 3.681 (2.4102) | 6.193 (6.3784) | 3.885 (2.7228) | 4.631 (3.7051) | 3.785 (3.2552)

7. Secondary Outcome: Terminal Rate Constant of Single Dose of Oxymorphone by Treatment Group
Description: λ: Terminal rate constant, calculated as the negative slope of the ln-linear portion of the terminal plasma concentration-time curve (single-dose period only)
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: Time -1
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | Single Dose of 6-OH-Oxymorphone: 10mg Tablet | Single Dose 6-OH-Oxymorphone: 15mg Tablet
Number analyzed (Participants) | 9 | 3 | 8 | 5 | 5 | 9
Time -1 | 0.209 (0.2552) | 0.214 (0.2962) | 0.073 (0.0549) | 0.281 (0.2072) | 0.101 (0.0965) | 0.042 (0.0234)

8. Secondary Outcome: Terminal Half-life of Single Dose of Oxymorphone by Treatment Group
Description: t½: Terminal half-life, calculated as terminal rate constant/(ln 2) (single-dose period only)
Time Frame: Baseline, 2h, 4h, 8h, 12h, 24h, 28h, 32h, 36h and 48h
Population: PK Population (only including subjects with sufficient evaluable time points for this outcome measure).
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Single Dose of 6-OH-Oxymorphone: 5mg Tablet | Single Dose of 6-OH-Oxymorphone: 10mg Tablet | Single Dose 6-OH-Oxymorphone: 15mg Tablet
Number analyzed (Participants) | 9 | 3 | 8 | 5 | 5 | 9
hour | 12.099 (9.9336) | 15.900 (18.2533) | 19.974 (22.4488) | 19.215 (37.3737) | 23.635 (33.6381) | 22.520 (15.3063)

ADVERSE EVENTS:
Time Frame: All AEs (Single Dose and Multiple Dose) were collected by the investigator starting 15 minutes after the first dose through the end of the study evaluation (24 hours post-first dose or early termination for Single Dose and 48 hours post first dose or early termination for Multiple Dose) and for up to 30 days after the last dose of study medication; this included any AEs that were ongoing at the completion/termination of the study.
Arm/Group | Single Dose of Oxymorphone IR: 5mg Tablet | Single Dose of Oxymorphone IR: 10mg Tablet | Single Dose of Oxymorphone IR: 15mg Tablet | Multiple Dose of Oxymorphone IR: 5mg Tablet | Multiple Dose of Oxymorphone IR: 10mg Tablet | Multiple Dose of Oxymorphone IR: 15mg Tablet
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/9 | 0/11 | 0/9 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 1/9 | 1/11 | 1/9 | 1/8 | 0/8
Other Adverse Events (participants affected / at risk) | 3/13 | 4/9 | 7/11 | 8/9 | 5/8 | 6/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose of Oxymorphone IR: 5mg Tablet (N=13) | Single Dose of Oxymorphone IR: 10mg Tablet (N=9) | Single Dose of Oxymorphone IR: 15mg Tablet (N=11) | Multiple Dose of Oxymorphone IR: 5mg Tablet (N=9) | Multiple Dose of Oxymorphone IR: 10mg Tablet (N=8) | Multiple Dose of Oxymorphone IR: 15mg Tablet (N=8)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fat embolism (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Failure of implant (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Pupils unequal (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0
Somatosensory evoked (Investigations) | 0 | 0 | 0 | 0 | 1 | 0
Monoplegia (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Spinal cord oedema (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Dose of Oxymorphone IR: 5mg Tablet (N=13) | Single Dose of Oxymorphone IR: 10mg Tablet (N=9) | Single Dose of Oxymorphone IR: 15mg Tablet (N=11) | Multiple Dose of Oxymorphone IR: 5mg Tablet (N=9) | Multiple Dose of Oxymorphone IR: 10mg Tablet (N=8) | Multiple Dose of Oxymorphone IR: 15mg Tablet (N=8)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 3
Tachycardia (Cardiac disorders) | 1 | 0 | 0 | 1 | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Constipation (Gastrointestinal disorders) | 1 | 0 | 1 | 3 | 4 | 1
Nausea (Gastrointestinal disorders) | 1 | 2 | 1 | 4 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1 | 0 | 2 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 4 | 1 | 0 | 2
Oxygen saturation decreased (Investigations) | 1 | 0 | 0 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 2 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 0 | 1 | 2 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 3 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 1 | 1 | 0 | 0 | 0 | 0
Sedation (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1 | 1 | 0
Urinary retention (Renal and urinary disorders) | 0 | 0 | 1 | 1 | 0 | 3
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 1 | 1

LIMITATIONS AND CAVEATS:
This post marketing study was required by the FDA. Endo Pharmaceuticals Inc. no longer promotes opioids and no longer markets Opana® ER.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No